CLINICAL TRIAL: NCT00952900
Title: An Implementation and Biobehavioral Study of TMJMD
Brief Title: An Implementation and Biobehavioral Study of Temporomandibular Joint and Muscle Disorder (TMJMD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Collaborators: Texas A&M University (Other)
Responsible Party: Principal Investigator, Robert J. Gatchel, Robert J. Gatchel, Ph.D., ABPP, Professor and Chair, Department of Psychology, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U01DE010713 (NIH); U01DE010713 (NIH)
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Temporomandibular Joint and Muscle Disorder
Keywords: TMJMD; Acute Pain; RDC/TMD; Community Treatment Clinics; RCT; Evidence-Based Outcomes; Short- and long-term follow-up; Biopsychosocial; Assessment and Treatment; Ability to read and write English; 6 months' or less duration of TMD; No other pain-related conditions
MeSH Terms: conditions — Muscular Diseases; Acute Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Early Biobehavioral Intervention (Experimental): This intervention involves the use of non-invasive treatment modalities such as relaxation/biofeedback, stress management, and cognitive coping skills. It is based upon previous clinical research studies demonstrating the efficacy of this intervention in allowing acute TMD patients to better cope with stress and lifestyle issues that produce the TMD pain/discomfort.
  Interventions: Behavioral: Biobehavioral
- Attention Control Group (Active Comparator): This intervention involves the presentation of helpful information to patients that explains etiology and potential treatment modalities used to modify/reduce TMD pain/discomfort.
  Interventions: Behavioral: Active Coping/Attention Intervention
- No Active Treatment Comparison Group (No Intervention): Unlike the other two treatment groups, that involve high-risk acute TMD patients, this group includes low-risk acute TMD patients. Past studies have shown that these low risk patients do not need any early intervention in order to prevent chronicity.

INTERVENTIONS:
Behavioral: Biobehavioral — 6 sessions of Biobehavioral treatment modalities that include relaxation/biofeedback, stress management, and coping skills techniques.
  Arms: Early Biobehavioral Intervention
Behavioral: Active Coping/Attention Intervention — 6 sessions of didactic educational techniques to expose patients to the causes of TMD, as well as introducing them to traditional treatment modalities for intervening with acute TMD problems.
  Arms: Attention Control Group

SUMMARY:
With the great economic costs and traditionally poor outcomes among chronic temporomandibular joint and muscle disorder (TMJMD) patients, it has become important to treat patients in the acute state, in order to prevent these more chronic disability problems. This has been the goal of two past funded grant projects. Results of the initial project isolated risk factors that successfully predicted the development of chronicity with a 91% accuracy rate. A statistical algorithm was developed which was used in the second project to screen out "high-risk" patients. These patients were then randomly assigned an early intervention or non-intervention group. One-year follow-up evaluations documented the treatment efficacy and cost effectiveness of early intervention. These results have major implications for effective early intervention and significant health care cost savings for this prevalent pain and disability problem. For the present proposed project, we plan to implement this treatment program in order to evaluate its effectiveness in more community-based dental practices. This is in response to NIH's request for the implementation of evidence-based treatment approaches, developed in controlled clinical settings, to the "real world" of diverse practices in the community. Acute TMJMD patients will be recruited from two community-based clinics. Based upon our "risk" screening algorithm, high-risk patients will be randomly assigned to one of two groups (n=225/group): an early biobehavioral intervention or an attention-control group. It is hypothesized that the attention control "high-risk" patients will display more chronic TMJMD problems, relative to the "high-risk" early intervention patients, at one- and two-year follow-ups. A number of biopsychosocial measures will be evaluated, including chewing performance, the RDC/TMD, self-reported pain and stress, etc. Such a multi-level, multi-systems approach has not been applied to better understand the biopsychosocial underpinnings of TMJMD. Results from this component of the project will greatly aid in stimulating future research leading to the better understanding of TMJMD, as well as better tailoring of prescribed treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Subject Must be an Adult Aged 18 or Older.
* Subject's First Acute Jaw Pain/Discomfort Episode Must Have First Developed Within the Last 6 Months

Exclusion Criteria:

* Younger than 18 years of age
* TMD pain/discomfort of greater than 6 months' duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2008-08; Primary Completion 2013-10 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Acute TMJMD does not progress to chronic | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Gatchel, Ph.D., ABPP, Principal Investigator — The University of Texas at Arlington
Locations (1):
- UT Arlington, Arlington, Texas, United States